CLINICAL TRIAL: NCT00609635
Title: The Association Between Cytokine Genotype Polymorphisms and Severity of RSV-Induced Illness in the Elderly
Brief Title: Association Between Cytokines and Severity of Respiratory Syncytial Virus (RSV)-Induced Illness in the Elderly
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: American Academy of Allergy, Asthma, and Immunology (Other)
Responsible Party: Ritu Pabby, MD, Allegheny General Hosptial Dept. of Allergy, Asthma, & Immunology
Other Study IDs: Adult RSV RC# 4212
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory; RSV-induced respiratory illness
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A buccal brushing (cells collected from the inside of the cheek) will be collected and stored for DNA analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
This research study involves studying the genes that may affect how ill you become during respiratory infection with respiratory syncytial virus (RSV). RSV is a virus that often causes common colds.

Cytokines are chemicals that are naturally made by your body. Cytokine levels are increased in some people when they have common colds or wheezing caused by respiratory syncytial virus (RSV). The purpose of this study is to study the genes that may control cytokine levels during infection with RSV in the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 65 years of age diagnosed with RSV-induced respiratory illness
* Diagnosis (based upon ICD-9-CM codes) for pneumonia, upper respiratory illness, bronchitis, COPD, asthma, viral illness, or congestive heart failure (CHF)
* Willing to sign informed consent.

Exclusion Criteria:

* Not willing to sign informed consent.
* Subjects less that 65 years of age
* Subjects not diagnosed with a respiratory illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: inpatient or outpatient subjects with respiratory illnesses potentially caused by RSV
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Pabby, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States